CLINICAL TRIAL: NCT04654013
Title: Effects of Near Vision Spectacle Correction on Work Retention Among Textile Factories Workers in India
Brief Title: PROductivity Study of Presbyopia Elimination in Rural-dwellers III
Acronym: PROSPERIII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: VisionSpring (Other); Clearly (Other); University of Michigan (Other); Good Business Lab (Unknown); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHLS 20_84
Record Dates: First submitted 2020-10-21; First posted 2020-12-04 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Presbyopia
Keywords: Presbyopia; Refractive error; Work retention; Spectacle wear compliance; Work efficiency
MeSH Terms: conditions — Presbyopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: 1260 workers aged 30 years and above with uncorrected presbyopia will be randomized to receive free glasses within one week of undergoing vision assessment, or free glasses at the end of the study assessment (18 months after vision assessment).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study personnel assessing trial outcomes will be masked as to participants assignment, which will be simplified by the fact that there will be participants with and without glasses at both Intervention and Control. It is not ethical in this setting to provide Control participants with placebo treatment (glasses with zero power lenses), but participants will not be informed of either the overall design of the study or the explicit treatment intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Workers assigned to the intervention group will receive free spectacles of a design they select, based on the worker's measured refractive power and dispensed one week later at the factory by the study ophthalmic personnel.
  Interventions: Device: Spectacles
- Control (No Intervention): Workers assigned to the Control group will receive similar free glasses at the end of the study assessment (18 months).

INTERVENTIONS:
Device: Spectacles — Intervention group workers receive free glasses within one week of undergoing vision assessment (May 2022). The duration of the treatment for the Intervention participants will depend on when they leave employment at the factor. If they stayed for the full duration of the trial, they will have undergone a maximum of 18 months (December 2023).
  Other Names: Eyeglasses; Reading glasses
  Arms: Intervention

SUMMARY:
The investigators will conduct an embedded mixed methods study in which the primary approach is a randomized controlled trial (RCT), and the secondary or embedded approach is a descriptive qualitative study. The aim of the RCT is to assess the impact of presbyopic correction on workplace productivity and retention in the textile industry in a low middle-income country. Additional qualitative data will be collected to enhance understanding of factors linked to reasons why enrolled sew-ers left their job during the study. Participants will be textile workers aged 30 years and above with uncorrected presbyopia who are employed by Shahi Exports Private Limited in Karnataka, India.

DETAILED DESCRIPTION:
Globally, 1.1 billion people lack a simple pair of reading glasses to correct impaired near vision, called presbyopia. Presbyopia can begin as early as age 30 years, commonly becomes functionally apparent by 40, and is essentially complete by 55 meaning that presbyopia is most common at the height of the working years. The global productivity loss due to uncorrected presbyopia has been estimated to exceed US$25 billion, and presbyopia is shown to be associated with significant impairment in activities of daily living. There is paucity in trial evidence of the impact on near vision spectacle correction on work productivity and workplace retention. The largest reported effect sizes among such trials (specifically for productivity) was the PROSPER trial, which showed that providing inexpensive near vision glasses increased the daily weight of tea picked among presbyopic, mostly-female Indian agricultural workers by more than 5 kg (21.7%) compared to those in the control group.

Study Plan: The investigators will choose 1260 textile workers aged 30 years and above with uncorrected presbyopia who are employed by Shahi Exports Private Limited in Karnataka, India. They will be randomly assigned into one of two groups: a group receiving free reading glasses within one week of undergoing vision assessment ("Intervention") or a group receiving identical reading glasses at the end of the assessment period ("Control").The main study outcome will be the proportion of workers who continue working at the factories in the intervention group (as opposed to control). The investigators anticipate that the glasses intervention will increase retention by 20% in the Intervention group at 1 year.

The study will also assess the workers' efficiency, why they have left employment, how satisfied and valued they felt at their work and how often they use their glasses for work. These other outcomes will help the investigators to better understand the causal pathway between vision and work retention. The investigators will also study the total cost of providing glasses per additional worker retain their employment.

Research question: Will providing free glasses to presbyopic Indian textile workers increase work retention?

Design: Investigator-masked, multi-center randomized controlled trial with a qualitative component

Rationale: Although presbyopia is safely, effectively and inexpensively treated with glasses, rates of optical correction in LMICs are as low as 10%. The way in which firms manage workers has profound implications for performance by way of worker attendance, retention, and productivity. Similarly, worker engagement, and the extent to which workers feel valued, is a key determinant of firm performance. As the low-skill workforce in many developing countries transitions rapidly from agriculture to industrial work, employers struggle with high worker turnover due to poor working conditions, low pay, and restricted worker rights. Few trials have been published which address the question of whether healthcare interventions can improve work performance as well as workplace retention, especially among persons over the age of 40 in low and middle-income countries (LMICs). There is interest in understanding if these results obtained in an agricultural setting can be extended to other financially-important sectors.

Methods: The investigators will choose 1260 textile workers aged 30 years and above with uncorrected presbyopia who are employed by Shahi Exports Private Limited in Karnataka, India. They will be randomly assigned into one of two groups: a group receiving free reading glasses within one week of undergoing vision assessment ("Intervention") or a group receiving identical reading glasses at the end of the assessment period ("Control").

The main outcome 18 month later will be work retention; secondary outcomes are workers' efficiency, the reasons the workers left their employment, satisfaction and perceived self-valued at work and glasses wear adherence at work. Attitudes about presbyopia and spectacle use and intervention cost-effectiveness will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years and above
* Distance visual acuity >= 6/12 in both eyes
* Presence of presbyopia, defined as the inability, correctable with reading glasses, to read the N8 line using both eyes together, on a tumbling near vision chart at a distance of 25cm, 30cm, 40cm, and 50cm based on workers working distance
* Employed at the factory for >=3months in the sewing department

Exclusion Criteria:

* Current ownership of reading or distance glasses (regardless of accuracy)
* Obvious evidence of ocular disease in either eye detected during the eye examination, or history of such disease based on self-report
* Low likelihood of completing follow-up in the study due to current plans to move out of the area or leave employment at Shahi during the follow-up period

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Work retention | September 2022 to May 2024; Over the 18 month follow-up period from enrolment to study completion
  Proportion of textile workers who continue to work at the textile factories assessed from trial entry to closure as recorded in Shahi's Human Resource Management Database

SECONDARY OUTCOMES:
Compliance with spectacle wear | 3, 6, 9, 12, 15 and 18 months after enrolment
  Actual presence of spectacles on the worker's face at work as reported by supervisor at the time of unannounced observation
Change in work satisfaction | Between baseline and 3, 6, 9, 12, 15 and 18 months after enrolment
  Proportion of sew-ers who state they are satisfied or very satisfied with work, feel valued or very valued at work, and are likely or very likely to stay with Shahi
Change in feeling valued-at-work | Between baseline and 3, 6, 9, 12, 15 and 18 months after enrolment
  Proportion of sew-ers who state they feel valued or very valued working at Shahi
Change in likeliness to stay at work | Between baseline and 3, 6, 9, 12, 15 and 18 months after enrolment
  Proportion of sew-ers who state they are likely or very likely to stay with Shahi
Change in work efficiency | Between baseline and 3, 6, 9, 12, 15 and 18 months after enrolment
  Self-assessed productivity scores using the Cantril's Ladder, with the best possible score being a 10, and the worst being a 0.
Attitudes towards vision correction | At month 0
  Worker's self-reported attitudes towards vision correction
Access to local eyecare services | At month 0
  Worker's self-reported access to local eyecare services
History of uptake of eyecare services | At month 0
  Worker's self-reported history of uptake of eyecare services
Change in Quality of Life as assessed by the THRIVE Near Vision Quality of Life tool | Between baseline and endline at 18 months
  Self-reported quality of life scores measured with the modified THRIVE Near Vision Quality of Life tool, a Likert Scale ranging from 1 (least affected) to 5 (worst affected).
Reasons leaving employment at Shahi | 2 months within participants leaving employment
  Reasons given by the former supervisor and colleagues of former sew-ers for workers no longer being employed at Shahi
Change in work productivity | Between baseline and 3, 6, 9, 12, 15 and 18 months after enrolment
  Proportion of target production realized by a worker per unit time.
Cost effectiveness of intervention | At study closeout at 18 months
  Ratio of incremental program cost to additional workers in the intervention group who retain employment vs. those in the control group. Incremental cost is the difference of program costs between implementation of intervention and control (not including study costs, such as data collection).
Change in skill grade | Between baseline and endline at 18 months
  Worker's skill grade as reported by supervisor.
Change in monthly wage | Between baseline and endline at 18 months
  Worker's monthly wage as reported by supervisor.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast
Locations (1):
- Good Business Lab, Bengaluru, Karantaka, India

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04654013/SAP_001.pdf